CLINICAL TRIAL: NCT05228093
Title: A Randomized Controlled Clinical Trial of Curative-intent Endoscopic Necrectomy Followed by Construction Using the Posterior Pedicle Nasal Septum and Floor Mucoperiosteum Flap Versus the Best Conservative Treatment for Mild and Moderate-grade Nasopharyngeal Necrosis
Brief Title: A Randomized Controlled Clinical Trial of Surgery Versus Conservative Treatment for Mild and Moderate-grade Nasopharyngeal Necrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Deputy director, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSFF-PRNN-2021
Record Dates: First submitted 2022-01-25; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Nasopharyngeal Carcinoma, Postradiation, Necrosis, Endoscopy Surgery, Conservative Treatment
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Necrosis | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery group (Experimental): Prior to surgery, a bacterial cultivation for purulent nasopharyngeal secretions and drug sensitivity assays were performed to identify sensitive antibiotics to be used postoperatively. Radical endoscopic necrectomy was performed under general anesthesia using the endoscopic endonasal approach. One side flap, typically the ipsilateral side, was harvested after complete radical endoscopic necrectomy.
  Interventions: Procedure: Curative-intent endoscopic necrectomy followed by reconstruction using the posterior pedicle nasal septum and floor mucoperiosteum flap
- Conservative group (Active Comparator): Patients receive debridement treatment of the necrotic tissues guided by endoscope and systematic antibiotic therapy partly under the guidance of nasopharyngeal secretion drug sensitivity test.
  Patients could use a common nasopharyngeal irrigation pot to wash the nasopharynx three times a day with warm boiled water or light saltwater (500 ml). If possible, patients could also received direct irrigation with an electronic nasopharyngoscopy operated by a physician.
  In addition, patients can receive hyperbaric oxygen therapy when conditions permit.
  Interventions: Procedure: Conservative treatment

INTERVENTIONS:
Procedure: Curative-intent endoscopic necrectomy followed by reconstruction using the posterior pedicle nasal septum and floor mucoperiosteum flap — Radical endoscopic necrectomy was performed under general anesthesia using the endoscopic endonasal approach. And the reconstruction of the nasopharyngeal defect use the nasal septum and floor mucoperiosteum flap. Antibiotic therapy based on the result of bacterial cultivation before the surgery was administered for 5-7 days after surgery. Patients are prescribed regional perfusion with recombinant human epidermal growth factor derivative liquid (Watsin Genetech Ltd, Shenzhen, Guangdong, P.R. China) to keep the wound humid, and endoscopic nasal cleanup was performed every 2-4 weeks until the flap was completely epithelialized and the entire defect was relined.
  Patients who were assessed as non-healing at 3 months after treatment will underwent salvage surgery.
  Arms: Surgery group
Procedure: Conservative treatment — Debridement guided by nasopharyngeal endoscopy and excision of the radiation-induced necrotic tissues were performed every 1 or 2 weeks. Patients are prescribed regional perfusion with recombinant human epidermal growth factor derivative liquid (Watsin Genetech Ltd, Shenzhen, Guangdong, P.R. China) to keep the wound humid. Other conservative treatment included daily nasopharynx rinsing with 2% aquae hydrogeniidioxide (5-10 mL each time) or saline (50-100 mL each time) and antibiotic therapy (metronidazole or ornidazole) guided by the culture results was also performed synchronously. Intravenous nutrition and systematic antibiotic therapy were also performed if indicated and necessary. In addition, patients can receive hyperbaric oxygen therapy when conditions permit.
  Patients who were assessed as non-healing at 3 months after treatment will underwent salvage surgery.
  Arms: Conservative group

SUMMARY:
Post radiation nasopharyngeal necrosis is a relatively special radiotherapy sequelae after radiotherapy for nasopharyngeal carcinoma. According to the degree of its development, it can be roughly divided into three stages: mild, moderate and severe stages, corresponding to the pre-nasopharyngeal necrosis stage, the soft tissue necrosis stage and the bone necrosis stage respectively. In the past, treatment methods were limited, including anti-infection, topical nasopharyngeal drugs, etc., the efficacy was not good, the nasopharyngeal necrosis lesions progressed, and a series of serious complications occurred, such as: intracranial infection secondary to osteonecrosis, massive nasopharyngeal hemorrhage, etc. It seriously endanger the life of the patient. With the continuous development of medical technology, the means of treatment are also constantly updated, such as repeated debridement guided by nasal endoscope, modified nasopharyngeal irrigation and hyperbaric oxygen therapy, the healing rate of nasopharyngeal necrosis has improved, especially the cure rate of patients in the mild and moderate-stages can reach 54.1%-54.8%. However, there are still some patients with poor healing of nasopharyngeal wounds after treatment.

Since 2004, our team has carried out a series of studies such as transnasal endoscopic nasopharyngeal resection combined with posterior pedicle nasal septum and floor mucoperiosteum flap(NSFF), and successfully achieved minimally invasive and en bloc resection of localized recurrent nasopharyngeal carcinoma. This method basically solved the problem of surgical wound healing of recurrent nasopharyngeal carcinoma. On this basis, we further applied it to the treatment of nasopharyngeal necrosis to further improve the cure rate and improve the prognosis. In addition, our retrospective study showed that compared with conservative treatment, curative-intent endoscopic necrectomy followed by reconstruction using the posterior pedicle nasal septum and floor mucoperiosteum flap can effectively prolong the overall survival time of patients and significantly improve the symptoms, but it still needs to be further confirmed by prospective clinical trials.

In addition, some patients (22.2%) had necrosis of the mucosal flap after receiving surgery, which affected the healing of surgical wounds. Besides, the development of nasopharyngeal necrosis is a slow process. If nasopharyngeal necrosis removal combined with pedicled mucosal flap repair is performed prematurely, the area outside the operation area may be necrotic again. Theoretically, each patient only has the nasal septum-nasal septum mucosal flaps on both sides of the nasal septum, which means that each patient only has 2 chances of repairing the nasal septum-nasal floor mucosal flaps. Premature surgical intervention may not only lead to incomplete debridement, but also lose a valuable opportunity for mucosal flap repair.

Therefore, based on the above problems, this study intends to compare the endoscopic nasopharyngeal necrosis debridement combined with pedicled mucosal flap repair versus the best conservative regimen for the treatment of early and mid-stage nasopharyngeal necrosis, to explore the prognosis of patients with nasopharyngeal necrosis. The preferred regimen, if confirmed by this study, is expected to standardize the treatment of nasopharyngeal necrosis after radiotherapy and further promote it, effectively increasing the cure rate of nasopharyngeal necrosis and improving the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Received radical radiotherapy for the nasopharynx;
2. For patients with early-stage and mid-stage nasopharyngeal necrosis diagnosed for the first time by clinical symptoms, imaging examinations and pathology. The lesions are limited to the superficial tissue of the nasopharynx and the deep tissue of each wall of the nasopharynx, regardless of the exposure of internal carotid artery invasion(ICA). For those patients with ICA exposure, vascular pretreatment (vascular embolization or bypass surgery) would be performed and reassess after 2-4 weeks of vascular treatment.
3. The patient has signed the informed notice and is willing and able to comply with the study plan visits, treatment plans, laboratory tests and other study procedures.

Exclusion Criteria:

1. Karnofsky score ≤ 70 points or Zubrod score > 2 points;
2. Patients with severe medical complications, insufficiency of important organs (heart, lung, liver, kidney) or neuropsychiatric disorders at the time of diagnosis.
3. Patients with pathologically confirmed local recurrence.
4. Cases who have received local nasal cavity and nasopharyngeal surgery in the past.
5. Patients who cannot cooperate with regular follow-up due to psychological, social, family and geographical reasons.
6. Other patients who are considered unsuitable for inclusion by the treating physician.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
The cure rate of nasopharyngeal necrosis at 3 months after enrollment | 3 months
  The cure rate of nasopharyngeal necrosis is defined as the complete re-epithelialization of the nasopharyngeal cavity, upon nasal endoscopic examination, and the mucosa; upon MRI examination.

SECONDARY OUTCOMES:
The Numeric Rating Scales (NRS) of pain | 3 months
  The Numeric Rating Scales (NRS) of pain was used to evaluate headaches level before and within 3 months after treatment. The patients were requested to rate their level of headache on a scale from 0 to 10, with 0 being none and 10 being unbearable.
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) overall | up to 1 year
  The quality of life was assessed per Quality of Life Questionnaire C30 (QLQ-C30).
Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) | up to 1 year
  The quality of life was assessed per Quality of Life Questionnaire Head and Neck Cancer-Specific Module (H&N35).
The cure rate of nasopharyngeal necrosis at 6 months after enrollment | 6 months
  Patients who was assessed as non-healing at 3 months after enrollment would receive salvage surgery. The cure rate of nasopharyngeal necrosis is reassessed at 3 months after salvage surgery.
Overall survival | up to 1 year
  The time from the date of randomization to the date of death due to any cause in an Intent-to-Treat analysis set.

CONTACTS AND LOCATIONS:
Overall Officials: Mingyuan Chen, MD, Principal Investigator — Sun Yat-sen University
Locations (4):
- China (4):
  - Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Hospital of Nanchang, Nanchang, Jiangxi